CLINICAL TRIAL: NCT04535141
Title: Addition of Olanzapine to Standard CINV Prophylaxis in Hematopoietic Stem Cell Transplant
Brief Title: Olanzapine for Nausea/Vomiting Prophylaxis in Recipients of Hematopoietic Stem Cell Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCCC2037; 20-0833 (Other: UNC Institutional Review Board)
Record Dates: First submitted 2020-08-18; First posted 2020-09-01 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Chemotherapy-induced Nausea and Vomiting; Chemotherapy; Nausea and Vomiting; Olanzapine
MeSH Terms: conditions — Vomiting; Nausea | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olanzapine Arm (Experimental): Olanzapine 5mg tablet with chemotherapy, and 3 days after
  Interventions: Drug: Olanzapine 5 MG
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine 5 MG — It will be a de-identified pill created by investigational drug services at University of North Carolina
  Other Names: Zyprexa
  Arms: Olanzapine Arm
Drug: Placebo — It will be a de-identified pill created by investigational drug services at University of North Carolina
  Arms: Placebo Arm

SUMMARY:
The purpose of this research study is to see if olanzapine helps to prevent nausea and/or vomiting (throwing up) when it is added to other medicines in subjects having stem cell transplants. Subjects will either be given olanzapine or an inactive pill (called a placebo) before getting any chemotherapy that is known to cause nausea and vomiting. During the study, the study coordinators will ask the subjects to complete surveys to understand if the patient is having nausea and vomiting, and if so, how bad it is making the patient feel.

This trial will split subjects into two groups: one group will be given an inactive pill (placebo), and the other group will be given the active pill (olanzapine). Study coordinators will collect surveys every morning before chemotherapy and 5 days after the last dose of chemotherapy. These surveys may be given by members of the study team or possibly on a mobile device.

Subjects may benefit from being in this research study because olanzapine may reduce the frequency or severity of chemotherapy-induced nausea and vomiting (CINV). The most common risks of using olanzapine include possibly becoming more tired, mild dizziness, mild low blood pressure, and mild muscle "quivering." Other possible adverse effects include low blood pressure, muscle weakness, increased appetite, weight gain, constipation, and liver function test changes however these risks are less common in subjects with cancer. In addition, there may be a change detected in heart rhythm however subjects will be screened for this ahead of time.

DETAILED DESCRIPTION:
Chemotherapy induced nausea and vomiting (CINV) occurs in up to 80% of patients on active therapy and remains a significant barrier to quality of life. CINV can alter electrolytes and enteral nutrition which can have a detrimental effect on patient adherence and health outcomes. Hematopoietic Stem Cell Transplant (HCT) patients are at increased risk for CINV because many of the conditioning regimens require multiple days of high-dose chemotherapy that are, in many cases, associated with highly-emetogenic potential.

Thus, most conditioning regimens require a 3-drug regimen for optimal CINV prophylaxis.

Current Standard of Care Current guidelines support the use of olanzapine in addition to a 3 drug CINV regimen for highly emetogenic chemotherapy, however some controversy remains as to olanzapine's place in therapy with moderately emetogenic chemotherapy. In HCT, current practice at University of North Carolina utilizes an neurokinin-1 receptor antagonist (NK1 RA), serotonin receptor antagonists (5-HT3 RA) and corticosteroid for CINV prophylaxis in conditioning regimens including moderate and highly emetogenic chemotherapy in accordance with American Society of Clinical Oncology (ASCO) and National Comprehensive Cancer Network (NCCN) recommendations.

Olanzapine, an atypical antipsychotic, antagonizes dopamine, serotonin, catecholamines, acetylcholine, and histamine receptors which helps prevent acute, breakthrough and delayed nausea. Olanzapine has shown benefit when used as prophylaxis in solid tumor patients receiving single-day highly emetogenic chemotherapy. The addition of olanzapine to 5HT-3 antagonist, NK-1 antagonist, and dexamethasone resulted in significantly more complete responses (CR) and more patients without CINV when compared to placebo in the acute, delayed and overall time periods. Data with olanzapine as CINV prophylaxis is not clear in HCT patients, but one retrospective study by Trifilio et. al. illustrates possible benefit in HCT. They compared an aprepitant-based regimen (aprepitant, ondansetron, and steroid) to an olanzapine-based regimen (olanzapine, ondansetron, and steroid) and found that patients in the olanzapine group had significantly less acute and delayed nausea. In addition, the olanzapine-based regimen required significantly less PRN rescue medication compared to the aprepitant based regimen. These results ultimately provided the foundation for the FOND-O study, a prospective trial that added olanzapine as part of CINV prophylaxis in both hematologic malignancies and HCT patients. The FOND-O study compared fosaprepitant, ondansetron, and dexamethasone (FOND) to fosaprepitant, ondansetron, dexamethasone and olanzapine (FOND-O). The inclusion of olanzapine resulted in significantly less delayed and overall nausea but did not affect the acute phase. While the FOND-O study was the first to look at utilizing olanzapine as part of 4 drug CINV prophylaxis in HCT, there were only 68 HCT patients included in the study. Only 24 allogeneic transplants and 44 autologous transplants were enrolled, and only 34 of these patients actually received olanzapine.

In addition, the FOND-O study utilized an olanzapine dose of 10 mg on each day of chemotherapy continued through chemotherapy day 3. Rationale for Clinical Study The purpose of our proposed study is to build upon the FOND-O results by doing a prospective, randomized, placebo-controlled study, focused entirely on HCT recipients, and powered to detect olanzapine's potential role in CINV prophylaxis in recipients of HCT. Based upon the available literature in both solid and hematologic malignancies the benefit outweighs the risk of adding olanzapine to standard CINV prophylaxis. The primary endpoint is complete response- defined as no emesis and no more than minimal nausea starting with the first dose of highly or moderately emetogenic conditioning chemotherapy and continuing 5 days beyond the last dose of highly or moderately emetogenic conditioning chemotherapy. Secondary endpoints are defined explicitly

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. Recipients receiving autologous or allogeneic HCT for any disease
3. Any conditioning chemotherapy regimen considered a standard bone marrow transplantation conditioning regimen
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
5. The subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

Exclusion Criteria:

1. Patients must not have started conditioning chemotherapy prior to consent. Note: test dose Busulfan is not part of conditioning chemotherapy
2. Known allergy to olanzapine
3. Baseline corrected QT interval ( QTc )>500 msec as calculated by the Fridericia formula
4. Patients receiving post-transplant cyclophosphamide as planned graft-versus-host disease (GVHD) prophylaxis
5. Pregnant or breastfeeding (NOTE: patients pregnant or breast-feeding are not eligible to proceed to transplant).
6. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
7. Treatment with any investigational drug within 7 days prior to registration.
8. Subject is receiving prohibited medications (ciprofloxacin or fluvoxamine) that cannot be discontinued/replaced by an alternative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ptachcinski, PharmD, Principal Investigator — jonathan.Ptachcinski@unchealth.unc.edu
Locations (1):
- UNC Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monson T, Greer D, Kreikemeier E, Liewer S. Olanzapine as a rescue antiemetic in hematopoietic stem cell transplant. J Oncol Pharm Pract. 2020 Jun;26(4):918-922. doi: 10.1177/1078155219879215. Epub 2019 Oct 21. PMID 31635549
- [Background] Navari RM, Qin R, Ruddy KJ, Liu H, Powell SF, Bajaj M, Dietrich L, Biggs D, Lafky JM, Loprinzi CL. Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Jul 14;375(2):134-42. doi: 10.1056/NEJMoa1515725. PMID 27410922
- [Background] Hesketh PJ, Kris MG, Basch E, Bohlke K, Barbour SY, Clark-Snow RA, Danso MA, Dennis K, Dupuis LL, Dusetzina SB, Eng C, Feyer PC, Jordan K, Noonan K, Sparacio D, Somerfield MR, Lyman GH. Antiemetics: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Oct 1;35(28):3240-3261. doi: 10.1200/JCO.2017.74.4789. Epub 2017 Jul 31. PMID 28759346
- [Background] Trifilio S, Welles C, Seeger K, Mehta S, Fishman M, McGowan K, Strejcek K, Eiten E, Pirotte C, Lucier E, DeFrates S, Mehta J. Olanzapine Reduces Chemotherapy-induced Nausea and Vomiting Compared With Aprepitant in Myeloma Patients Receiving High-dose Melphalan Before Stem Cell Transplantation: A Retrospective Study. Clin Lymphoma Myeloma Leuk. 2017 Sep;17(9):584-589. doi: 10.1016/j.clml.2017.06.012. Epub 2017 Jun 20. PMID 28694084
- [Background] Navari RM, Aapro M. Antiemetic Prophylaxis for Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Apr 7;374(14):1356-67. doi: 10.1056/NEJMra1515442. No abstract available. PMID 27050207
- [Background] Clemmons AB, Orr J, Andrick B, Gandhi A, Sportes C, DeRemer D. Randomized, Placebo-Controlled, Phase III Trial of Fosaprepitant, Ondansetron, Dexamethasone (FOND) Versus FOND Plus Olanzapine (FOND-O) for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Patients with Hematologic Malignancies Receiving Highly Emetogenic Chemotherapy and Hematopoietic Cell Transplantation Regimens: The FOND-O Trial. Biol Blood Marrow Transplant. 2018 Oct;24(10):2065-2071. doi: 10.1016/j.bbmt.2018.06.005. Epub 2018 Jun 13. PMID 29906570
- [Background] Basch E, Dueck AC, Rogak LJ, Mitchell SA, Minasian LM, Denicoff AM, Wind JK, Shaw MC, Heon N, Shi Q, Ginos B, Nelson GD, Meyers JP, Chang GJ, Mamon HJ, Weiser MR, Kolevska T, Reeve BB, Bruner DW, Schrag D. Feasibility of Implementing the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events in a Multicenter Trial: NCCTG N1048. J Clin Oncol. 2018 Sep 11;36(31):JCO2018788620. doi: 10.1200/JCO.2018.78.8620. Online ahead of print. PMID 30204536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 08/18/2020 through 03/17/2022 at 1 cancer center in North Carolina.
Pre-assignment Details: A total of ninety-four participants consented and three subjects withdrew their consent, and ninety-one enrolled in the study.
Groups:
- Usual Care: All subjects received the usual care and did not receive olanzapine.
- Olanzapine: All subjects received both olanzapine and usual care.
Period: Overall Study
Arm/Group | Usual Care | Olanzapine
Started | 46 | 45
Completed | 46 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Olanzapine | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 56
  >=65 years | 17 | 18 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 23 | 28 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 42 | 40 | 82
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 14 | 22
  White | 34 | 25 | 59
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: The number of subjects who completed the study and the overall rate of complete response were assessed.
  Complete response achievement requires all three of the following criteria for the entire duration of the study assessment period: 1. No emesis, 2. Response to PRO-CTCAE question "In the last 24 hours, how often did you have nausea?" is no higher than rarely and 3. Response to PRO-CTCAE question "In the last 24 hours, what was the severity of your nausea at its worst? a score no higher than "mild".
Time Frame: End of study assessment period, until 5 days after last chemotherapy administration (2- 12 days)
Population: The participants enrolled in the study and complete responses were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  The number of participants achieved a complete response | 13 | 21
  The number of participants did not achieve a complete response | 33 | 24

2. Secondary Outcome: Total Number of Rescue Medications Needed Acute
Description: The total number of rescue medications needed acute was calculated, starting from the first dose of highly or moderately emetogenic conditioning chemotherapy and continuing for one day after the last dose of highly or moderately emetogenic conditioning chemotherapy.
  The rescue medication is defined as documented administration of an anti-emetic agent other than those that are scheduled for chemotherapy-induced nausea and vomiting (CINV) prophylaxis.
Time Frame: End of day 1 following last chemotherapy administration. (Up to day 2)
Population: The subjects who completed CINV prophylaxis treatment and their rescue medications were counted.
Measure: Mean (Full Range); unit: number of rescue medication
Groups:
- Usual Care: All subjects who received the usual care and did not receive olanzapine.
- Olanzapin: All subjects received both olanzapine and usual care.
Arm/Group | Usual Care | Olanzapin
Number analyzed (Participants) | 46 | 45
number of rescue medication | 0.08 [0 to 2] | 0.10 [0 to 2]

3. Secondary Outcome: Number of Subjects Achieving Minimal Nausea
Description: To determine the number of subjects achieving minimal nausea was defined as the frequency of participants responded to the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) nausea question "In the last 24 hours, how often did you have nausea?" as "rarely or less" Starting with the first dose of chemotherapy and continuing for one day after the last dose of highly or moderately emetogenic conditioning chemotherapy.
  PRO-CTCAE of nausea scale includes categories: Never, Rarely, Occasionally, Frequently, Almost constantly To meet this endpoint the score reported for the Pro-CTCAE question for nausea frequency cannot exceed "rarely" and the score reported for the Pro-CTCAE question for nausea severity cannot exceed "mild"
Time Frame: Day 2-12
Population: The subjects who completed CINV prophylaxis treatment and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: All subjects who received the usual care, and did not receive olanzapine.
- Olanzapine: All subjects received both the usual care and olanzapine.
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  Yes | 15 | 25
  No | 31 | 20

4. Secondary Outcome: Frequency of Nausea in the Acute Phase
Description: Starting with the first dose of highly or moderately emetogenic conditioning chemotherapy and continuing for one day after the last dose of highly or moderately emetogenic conditioning chemotherapy.
  Nausea was assessed using subjects' responses to the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) nausea questions. Scale: Never, Rarely, Occasionally, Frequently, Almost constantly.
  To meet this endpoint the score reported for the Pro-CTCAE question for nausea frequency cannot exceed "rarely" in the first 24 hours following receipt of chemotherapy.
Time Frame: End of day 1 following last chemotherapy administration (Up to day 2)
Population: The subjects who completed CINV prophylaxis acute phase and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  Met endpoint | 43 | 44
  Did not meet endpoint | 3 | 1

5. Secondary Outcome: Number of Subjects Achieved Emesis Endpoint in Acute Phase.
Description: : The number of subjects who did not experience emesis, starting from the first dose of highly or moderately emetogenic conditioning chemotherapy and continuing for one day after the last dose of highly or moderately emetogenic conditioning chemotherapy. Met endpoint = 0 emesis.
Time Frame: End of day 1 following last chemotherapy administration. (Up to day 2)
Population: The subjects who completed CINV prophylaxis acute phase and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  Met endpoint | 45 | 45
  Did not meet endpoint | 1 | 0

6. Secondary Outcome: Frequency of Somnolence
Description: The frequency of somnolence was determined as the number of patients who experienced somnolence based on Common Terminology Criteria for Adverse Events version 5 (CTCAE v5). The number of subjects has somnolence during the study period was counted.
Time Frame: Day 2-12
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 43
Participants
  subjects have somnolence | 0 | 1
  subjects do not have somnolence | 46 | 42

7. Secondary Outcome: Safety Endpoint: Qtc Prolongation
Description: Prolongation of corrected QTc interval graded as defined in Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Corrected QTc was calculated using Fredericia's Formula. Corrected QT interval (QTc) = QT interval / (60/Heart rate)^0.33.
Time Frame: Day 1 to 5 days after end of the chemotherapy (Days 2- 12).
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Usual Care: All subjects received the usual care and did not receive olanzapine. EKG was performed at baseline.
- Baseline Olanzapine: All subjects received both olanzapine and usual care. EKG was performed at baseline.
- Usual Care Post-chemo Day 1: All subjects received the usual care and did not receive olanzapine. EKG was performed on post-chemo day 1
- Olanzapine Post-chemo Day 1: All subjects received both olanzapine and usual care. EKG was performed at post-chemo day 1
- Usual Care End of Study: All subjects received the usual care and did not receive olanzapine. EKG was performed at the end of the study
- Olanzapine- End of Study: All subjects received both olanzapine and usual care. EKG was performed at end of study
Arm/Group | Baseline Usual Care | Baseline Olanzapine | Usual Care Post-chemo Day 1 | Olanzapine Post-chemo Day 1 | Usual Care End of Study | Olanzapine- End of Study
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 46 | 45
Participants
  Grade 1 | 3 | 4 | 2 | 3 | 3 | 3
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0
  None | 43 | 41 | 44 | 42 | 42 | 41

8. Secondary Outcome: Number of Subjects Achieved Nausea Endpoint in the Delayed Phase.
Description: Nausea was assessed using subjects' responses to the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) nausea questions, starting the second day after the completion of highly or moderately emetogenic conditioning chemotherapy and continuing through the fifth day after the completion of highly or moderately emetogenic chemotherapy.
  Scale: Never, Rarely, Occasionally, Frequently, Almost constantly.
  The number of subjects who experienced "never" or "rarely" nausea were considered as met the endpoint while those who experienced "occasionally", "frequently" or "almost constantly" were considered as not met the endpoint.
Time Frame: Day 1 to 5 days after end of the chemotherapy (Days 2-12).
Population: The subjects who completed the treatment and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  Met endpoint | 19 | 27
  Did not meet endpoint | 27 | 18

9. Secondary Outcome: Severity of Nausea in Delayed Phase
Description: The severity of nausea in the delayed phase was defined as the response of the subject to the PRO- CTCAE nausea question.
  Starting the second day after the completion of highly or moderately emetogenic conditioning chemotherapy and continuing through the fifth day after the completion of highly or moderately emetogenic chemotherapy (PRO-CTCAE) Scale: Never, Rarely, Occasionally, Frequently, Almost constantly
  o meet the endpoint, the subject could not have answered a score as higher than "mild" in the period of time starting 24 hours after the last dose of chemotherapy and continuing until the 5th day following receipt of chemotherapy .
Time Frame: Day 2-12
Population: The subjects who completed the treatment and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  Met endpoint | 23 | 31
  Did not meet endpoint | 23 | 24

10. Secondary Outcome: Number of Emesis Episodes in Delayed Phase
Description: The number of emesis episodes in acute phase was defined as the number of subjects with no emesis, 1 emesis, and 2 or more emesis.
Time Frame: Day 1 to 5 days after end of the chemotherapy ( Days 2-12).
Population: The subjects who completed the treatment and responded to PRO-CTCAE questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
Participants
  No emesis episodes | 32 | 36
  1 emesis episode | 9 | 6
  2 or more emesis episodes | 5 | 3

11. Secondary Outcome: Total Number of Rescue Medications Needed -Delayed
Description: The total number of rescue medications needed for breakthrough chemotherapy-induced nausea and vomiting were calculated, starting from the second day after the completion of highly or moderately emetogenic conditioning chemotherapy and continuing through the fifth day after the completion of highly or moderately emetogenic chemotherapy.
  The rescue medication is defined as documented administration of an anti-emetic agent other than those that are scheduled for CINV prophylaxis.
Time Frame: Day 1 to 5 days after end of the chemotherapy ( Days 2-12).
Population: The subjects who completed CINV prophylaxis treatment and their rescue medications were counted.
Measure: Mean (Full Range); unit: number of rescue medication
Arm/Group | Usual Care | Olanzapine
Number analyzed (Participants) | 46 | 45
number of rescue medication | 0.47 [0 to 44] | 1.17 [0 to 22]

ADVERSE EVENTS:
Time Frame: from the first day of the study treatment until end of the treatment (Up to 24 days)
Description: Adverse events were assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0, from the first day of the study to the end of the treatment.
Arm/Group | Usual Care | Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/46 | 8/45
Other Adverse Events (participants affected / at risk) | 46/46 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=46) | Olanzapine (N=45)
Arrhythmia (Cardiac disorders) | 2 | 0
engraftment syndrome (Immune system disorders) | 1 | 4
Encephalopathy (Nervous system disorders) | 0 | 1
cytokine release syndrome (Immune system disorders) | 0 | 1
Syncopal episode (General disorders) | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=46) | Olanzapine (N=45)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 14 | 11
Akathisia (Nervous system disorders) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 3
Chest pain (General disorders) | 1 | 0
Confusion (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 20 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine increase (Investigations) | 2 | 3
Depression (Nervous system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 16 | 19
Dizziness (Nervous system disorders) | 3 | 0
Dry skin (Nervous system disorders) | 0 | 1
Dysgeusia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Ear and labrynth disorder (Ear and labyrinth disorders) | 0 | 1
Elevated alkaline phosphatase (Investigations) | 1 | 1
Alanine transaminase elevated (Investigations) | 1 | 1
aspartate aminotransferase elevated (Investigations) | 1 | 5
hyperglycemia (Metabolism and nutrition disorders) | 9 | 8
blood bilirubin increased (Investigations) | 1 | 0
Extrapyramidal symptom (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
fever (General disorders) | 0 | 1
Headache (Nervous system disorders) | 10 | 7
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hot flashes (Vascular disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 9 | 7
Hyperuricemia (Renal and urinary disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
anxiety (Psychiatric disorders) | 0 | 1
Infection (Infections and infestations) | 2 | 1
Insomnia (Psychiatric disorders) | 6 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 3 — mood change
Mucositis (Gastrointestinal disorders) | 0 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 2 — Other electrolyte abnormality
Pain (General disorders) | 5 | 5
Parkinsonian symptom (Nervous system disorders) | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
subconjunctival hemorrhage (Eye disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 13 | 4
Syncope (Cardiac disorders) | 1 | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Blood and lymphatic system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Xerostomia (Endocrine disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT04535141/Prot_SAP_000.pdf